CLINICAL TRIAL: NCT03905525
Title: A 48-week, 6-arm, Randomized, Double-blind, Placebo-controlled Multicenter Trial to Assess the Safety and Efficacy of Multiple CFZ533 Doses Administered Subcutaneously in Two Distinct Populations of Patients With Sjogren's Syndrome (TWINSS)
Brief Title: Study of Safety and Efficacy of Multiple Doses of CFZ533 in Two Distinct Populations of Patients With Sjogren's Syndrome
Acronym: TWINSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCFZ533B2201; 2018-004476-35 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-04-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Sjögren Syndrome
Keywords: Sjögren; fatigue; dryness; anti-CD40; CFZ533; iscalimab; TWINSS; autoimmune
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue | interventions — iscalimab

STUDY DESIGN:
Intervention Model Description: Patients will be screened and enrolled into one of the 2 study Cohorts:
  Cohort 1: At baseline subjects will be randomized in ratio 1:1:1:1 into one of three CFZ533 (iscalimab) arms (A, B or C) or to placebo (Arm D). After completion of 24 weeks of treatment (Period 1) placebo patients (Arm D) will be switched to active treatment (Arm D1) for the subsequent 24 weeks (Period 2).
  Cohort 2: At baseline subjects will be randomized in ratio 1:1 to iscalimab (Arm E) or to placebo (Arm F). After completion of 24 weeks of treatment (Period 1), placebo patients (Arm F) will be switched to iscalimab active treatment (Arm F1) for the subsequent 24 weeks (Period 2).
  All patients treated with iscalimab (Arms A,B,C,and E) in Period 1 will continue the same study treatment in Period 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, investigator staff, persons performing the assessments, will remain blind to the identity of the treatment within each cohort from the time of randomization until end of the study visit (week 60)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 /Arm A (Experimental): CFZ533 dose 1
  Interventions: Drug: CFZ533
- Cohort 1/Arm B (Experimental): CFZ533 dose 2
  Interventions: Drug: CFZ533
- Cohort 1/Arm C (Experimental): CFZ533 dose 3
  Interventions: Drug: CFZ533
- Cohort 1/Arm D (Placebo Comparator): Placebo dose (up to week 24)
  Interventions: Other: Placebo
- Cohort 1/Arm D1 (Experimental): CFZ533 dose 1 (from week 24)
  Interventions: Drug: CFZ533
- Cohort 2/Arm E (Experimental): CFZ533 dose 1
  Interventions: Drug: CFZ533
- Cohort 2/Arm F (Placebo Comparator): Placebo dose (up to week 24)
  Interventions: Other: Placebo
- Cohort 2/Arm F1 (Experimental): CFZ533 dose 2 (from week 24)
  Interventions: Drug: CFZ533

INTERVENTIONS:
Drug: CFZ533 — Biological
  Other Names: iscalimab
  Arms: Cohort 1 /Arm A; Cohort 1/Arm B; Cohort 1/Arm C; Cohort 1/Arm D1; Cohort 2/Arm E; Cohort 2/Arm F1
Other: Placebo — liquid placebo for injections
  Arms: Cohort 1/Arm D; Cohort 2/Arm F

SUMMARY:
This study will evaluate safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple doses of CFZ533 (iscalimab) in patients with Sjögren's Syndrome.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multicenter study of CFZ533 in 2 distinct populations (cohorts) of patients with Sjögren's Syndrome: 1) moderate-to-severe disease (systemic and symptomatic involvement) and; 2) low systemic involvement but high symptom burden.

The study includes up to 6 weeks screening period, 48 weeks of treatment (divided into treatment periods of 24 weeks each) and 12 weeks follow up. Study treatment will be administered as bi-weekly subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female patient ≥ 18 years of age
* Classification of Sjögren's Syndrome according to ACR/EULAR 2016 criteria (Shiboski et al 2017)
* Seropositive for anti-Ro/SSA antibodies
* Stimulated whole salivary flow rate of ≥ 0.1 mL/min

Inclusion criteria specific for Cohort 1:

* ESSDAI ≥ 5 within the 8 predefined organ domains
* ESSPRI score of ≥5

Inclusion criteria specific for Cohort 2:

* ESSDAI < 5 within 8 domains scored for inclusion criterion for Cohort 1
* ESSPRI fatigue subscore ≥ 5 or ESSPRI dryness subscore ≥ 5

Exclusion Criteria:

* Sjögren's Syndrome overlap syndromes where another autoimmune rheumatic disease constitutes the principle illness
* Use of other investigational drugs
* Prior use of B cell depleting therapies, abatacept or any other immunosuppressants unless specifically allowed be the protocol.
* Use of steroids at dose >10 mg/day.
* Uncontrolled ocular rosacea (affecting the eye adnexa), posterior blepharitis or Meibomian gland disease (this criterion applies only to patients considered for Cohort 2)
* Active viral, bacterial or other infections requiring systemic treatment
* Receipt of live/attenuated vaccine within a 2-month period prior to randomization.
* Chronic infection with hepatitis B (HBV) or hepatitis C (HCV).
* Evidence of active tuberculosis (TB) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Change in EULAR Sjögren Syndrome Disease Activity Index (ESSDAI) score from baseline at 24 weeks as compared to placebo | 24 weeks
  Cohort 1 - Efficacy
Change in EULAR Sjögren Syndrome Patient Reported Index (ESSPRI) score from baseline at 24 weeks as compared to placebo. | 24 weeks
  Cohort 2 - Efficacy

SECONDARY OUTCOMES:
Change from baseline in ESSPRI at Week 24 | 24 weeks
  Cohort 1 - Efficacy (Patient Reported Outcomes)
Change from baseline in score of Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire at Week 24 | 24 weeks
  Cohort 1&2 - Efficacy (Patient Reported Outcomes)
Change from baseline in Physician Global Assessment (PhGA) at Week 24 | 24 weeks
  Cohort 1&2 - Efficacy (Clinical Outcome Measures)
Change from baseline in ESSDAI at Week 24 | 24 weeks
  Cohort 2 - Efficacy (Clinical Outcome Measures)
Proportion of subjects with at least 12 points improvement measured by score of Impact of Dry Eye on Everyday Life (IDEEL) questionnaire symptom bother module at Week 24. | 24 weeks
  Cohort 2 - Efficacy (Patient Reported Outcomes)
Incidence of adverse events (AEs), serious adverse events (SAEs) from baseline to Week 24 and from week 24 to the end of study | 60 weeks
  Cohort 1&2 - Safety
Serum Free Light Chain (FLC) levels at analysis visit up to end of study | 60 weeks
  Cohort 1&2 - Biomarkers (1)
Immunoglobulin IgG and IgM levels at analysis visits up to end of study | 60 weeks
  Cohort 1&2 - Biomarkers (2)
Percent change from baseline in plasma CXCL-13 levels at analysis visits up to end of study | 60 weeks
  Cohort 1&2 - Biomarkers (3)
  Chemokine (C-X-C motif) ligand 13 (CXCL13), also known as B lymphocyte chemoattractant (BLC) or B cell-attracting chemokine 1 (BCA-1), is a protein ligand that in humans is encoded by the CXCL13 gene.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (69):
- United States (8):
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Madison, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, CABA
- Novartis Investigative Site, Nedlands, Western Australia, Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Brazil (3):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (4):
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Concepción
  - Novartis Investigative Site, Santiago
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Cali, Valle del Cauca Department
- France (5):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (4):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Athens, Greece
- Hungary (3):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Udine, UD
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Portugal (3):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
- Romania (2):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
- Russia (6):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Novartis Investigative Site, Stockholm, SE, Sweden
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fisher BA, Mariette X, Papas A, Grader-Beck T, Bootsma H, Ng WF, van Daele PLA, Finzel S, Noaiseh G, Elgueta S, Hermann J, McCoy SS, Akpek E, Bookman A, Sopala M, Montecchi-Palmer M, Luo WL, Scheurer C, Hueber W; TWINSS study group. Safety and efficacy of subcutaneous iscalimab (CFZ533) in two distinct populations of patients with Sjogren's disease (TWINSS): week 24 results of a randomised, double-blind, placebo-controlled, phase 2b dose-ranging study. Lancet. 2024 Aug 10;404(10452):540-553. doi: 10.1016/S0140-6736(24)01211-X. Epub 2024 Jul 31. PMID 39096929